CLINICAL TRIAL: NCT04537949
Title: A Multi-site, Phase I/II, 2-Part, Dose-Escalation Trial Investigating the Safety and Immunogenicity of a Prophylactic SARS-CoV-2 RNA Vaccine (BNT162b3) Against COVID-19 Using Different Dosing Regimens in Healthy Adults
Brief Title: A Trial Investigating the Safety and Effects of One BNT162 Vaccine Against COVID-19 in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BNT162-04; 2020-003267-26 (EudraCT Number); U1111-1254-4840 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2020-09-02; First posted 2020-09-03 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Covid-19; Protection Against COVID-19
Keywords: Protection against COVID-19; Coronavirus; Vaccine; RNA Vaccine; SARS-CoV-2; Coronavirus Disease 2019; Virus Diseases; Coronavirus infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A participants aged 18 to 55 years (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b3
- Part A participants aged 56 to 85 years (optional) (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b3

INTERVENTIONS:
Biological: BNT162b3 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime/Boost (P/B) regimen).

SUMMARY:
Originally, the study was planned to include two parts, i.e., Part A and Part B, however Part B was skipped due to changes in the overall clinical development plan. The conducted Part A was a dose-finding part to investigate the optimal dose, allowing dose adjustments upwards and downwards in younger participants. Doses tested in older participants were chosen based on acceptability of dosing in younger participants.

DETAILED DESCRIPTION:
This study was a multi-site, Phase I/II, open-label, dose-escalation study. The study included the first in human dose and dose ranging groups in healthy younger participants (aged 18 to 55 years [yrs]) and older participants (aged 56 to 85 yrs). The conducted Part A followed a dose escalation design. Discretionary dose de-escalation and refinement was also planned. Study participants with the first-in-human [FIH] immunization and any subsequent dose escalation cohorts were immunized using a sentinel dosing/subject staggering. For any dose de-escalation or dose-refinement cohorts in younger adults, i.e., cohorts with doses lower than previously tested, participants were dosed using a subject staggering process. Cohorts in older participants were optional and dependent on acceptability of dosing in younger participants. Part A consisted of a treatment phase (screening to Visit 7) and a follow-up phase (Visits 8 to 10).

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent by signing the informed consent form (ICF) before initiation of any trial-specific procedures.
* They must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (e.g., to practice social distancing and to follow good practices to reduce their chances of being infected or spreading COVID-19), and other requirements of the trial.
* They must be able to understand and follow trial-related instructions.
* For younger adult cohorts, volunteers must be aged 18 to 55 years, have a body mass index over 19 kg/m^2 and under 30 kg/m^2 (i.e., be neither underweight nor obese), and weigh at least 50 kg at Visit 0.

OR For older adult cohorts, volunteers must be aged 56 to 85 years, have a body mass index over 19 kg/m^2 and under 30 kg/m^2 (i.e., be neither underweight nor obese), and weigh at least 50 kg at Visit 0.

* They must be healthy, in the clinical judgment of the investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs (systolic/diastolic blood pressure, pulse rate, body temperature, respiratory rate), and clinical laboratory tests (blood chemistry, hematology, and urine chemistry) at Visit 0.
* Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin urine test at Visit 0 and Visit 1. Women that are postmenopausal or permanently sterilized will be considered as not having reproductive potential.
* WOCBP must agree to practice a highly effective form of contraception during the trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization. WOCBP must agree to require their male partners to use condoms during sexual contact (unless male partners are sterilized or infertile).
* WOCBP must confirm that they practiced at least one highly effective form of contraception for the 14 days prior to Visit 0.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice a highly effective form of contraception with their female partner of childbearing potential during the trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* Men must be willing to refrain from sperm donation, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* They must have confirmation of their health insurance coverage prior to Visit 0.
* They must agree to not be vaccinated during the trial, starting after Visit 0 and continuously until 28 days after receiving the last immunization.

Exclusion Criteria:

* Have had any acute illness, as determined by the investigator, with or without fever, within 72 hours prior to the first immunization. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their well-being if they participate as trial participants in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Are breastfeeding on the day of Visit 0 or who plan to breastfeed during the trial, starting after Visit 0 and continuously until at least 90 days after receiving the last immunization.
* Have a known allergy, hypersensitivity, or intolerance to the planned investigational medicinal product (IMP) including any excipients of the IMP.
* Had any medical condition or any major surgery (e.g., requiring general anesthesia) within the past 5 years which, in the opinion of the investigator, could compromise their well-being if they participate as trial participants in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have any surgery planned during the trial, starting after Visit 0 and continuously until at least 90 days after receiving the last immunization.
* Had any chronic use (more than 21 continuous days) of any systemic medications, including immunosuppressants or other immune-modifying drugs, within the 6 months prior to Visit 0 unless in the opinion of the investigator, the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise participant safety.
* Received any vaccination within the 28 days prior to Visit 0.
* Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Visit 0.
* Had administration of another IMP including vaccines within 60 days or 5 half-lives (whichever is longer), prior to Visit 0.
* Have a known history or a positive test of any of human immunodeficiency virus (HIV) 1 or 2, Hepatitis B, or Hepatitis C, within the 30 days prior to Visit 0.
* Have a positive polymerase chain reaction (PCR)-based test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within the 30 days prior to Visit 1.
* Have a positive drugs of abuse (for amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, and tricyclic antidepressants) result at Visit 0 or Visit 1.
* Have a positive breath alcohol test at Visit 0 or Visit 1.
* Previously participated in an investigational trial involving lipid nanoparticles.
* Are subject to exclusion periods from other investigational trials or simultaneous participation in another clinical trial.
* Have any affiliation with the trial site (e.g., are close relative of the investigator or dependent person, such as an employee or student of the trial site).
* Have a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their well-being if they participate as trial participants in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have a history of hypersensitivity or serious reactions to previous vaccinations.
* Have a history of Guillain-Barré Syndrome within 6 weeks following a previous vaccination.
* Have a history of narcolepsy.
* Have history of alcohol abuse or drug addiction within 1 year before Visit 0.
* Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Visit 0.
* Have any abnormality or permanent body art (e.g., tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site.
* Have had any blood loss >450 mL, e.g., due to donation of blood or blood products or injury, within the 7 days prior to Visit 0 or plan to donate blood during the trial, starting after Visit 0 and continuously until at least 7 days after receiving the last immunization.
* Symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
* Have had contact with persons diagnosed with COVID-19 or who tested positive for SARS-CoV-2 by any diagnostic test within the 30 days prior to Visit 1.
* Are soldiers, participants in detention, contract research organization (CRO) or sponsor staff or their family members.
* Regular receipt of inhaled/nebulized corticosteroids.
* Have a condition known to put them at high risk for severe COVID-19, including those with any of the following risk factors:

  * Cancer
  * COPD (chronic obstructive pulmonary disease)
  * Immunocompromised state (weakened immune system) from solid organ transplant
  * Obesity (BMI of 30 or higher)
  * Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
  * Sickle cell disease
  * Diabetes mellitus
  * Hypertension
  * Asthma
  * Chronic liver disease
  * Known Stage 3 or worse chronic kidney disease (glomerular filtration rate <60 mL/min/1.73 m^2)
  * Anticipating the need for immunosuppressive treatment within the next 6 months
  * Resident in a long-term facility
  * Current vaping or smoking (occasional smoking is acceptable)
  * History of chronic smoking within the prior year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (2):
- Germany (2):
  - Contract Research Organization, Berlin
  - Contract Research Organization, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogel AB, Lui BG, Tompkins K, Kanevsky I, Muik A, Krumm SA, Guler A, Maddur MS, Walzer KC, Witzel S, Vascotto F, Stanganello E, Ota-Setlik A, Cottingham KJ, Allbritton O, Keverne J, Aragao-Santiago L, Swanson KA, Tureci O, Sahin U. Strong and early immune responses against SARS-CoV-2 in mice and rhesus macaques after BNT162b3 vaccination. NPJ Vaccines. 2026 Jan 13;11(1):10. doi: 10.1038/s41541-025-01365-w. PMID 41530185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were selected from the volunteer panel at the clinical CRO, volunteers who responded to either generic or study-specific advertisements in social media, or volunteers who contacted the clinical CRO via a web-based study participant recruitment portal. Study participants were selected from this pool of volunteers according to inclusion and exclusion criteria. The first participant was enrolled on 09 Sep 2020. The last visit of the last participant was on 07 Feb 2022.
Pre-assignment Details: All enrolled participants were allocated to treatment.
Groups:
- Part A Participants Aged 18 to 55 Years - 3 μg; Part A Participants Aged 18 to 55 Years - 10 μg; Part A Participants Aged 18 to 55 Years - 20 μg; Part A Participants Aged 56 to 85 Years - 3 μg; Part A Participants Aged 56 to 85 Years - 10 μg; Part A Participants Aged 56 to 85 Years - 20 μg; Part A Participants Aged 56 to 85 Years - 30 μg: BNT162b3: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime/Boost [P/B] regimen)
- Part A Participants Aged 18 to 55 Years - 30 μg: BNT162b3: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only, as decided by the Safety Review Committee).
Period: Treatment Phase
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — personal reasons not related to the IMP | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Phase
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Started | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 8 | 8 | 12 | 9 | 9 | 11 | 7 | 6
Not Completed | 3 | 4 | 0 | 3 | 3 | 1 | 5 | 6
Not completed — Roll-over into trial BNT162-14 | 3 | 1 | 0 | 2 | 1 | 1 | 5 | 6
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — personal reasons | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.32 (9.79) | 31.20 (9.11) | 31.89 (13.51) | 37.28 (6.40) | 66.08 (7.16) | 69.32 (8.74) | 64.93 (6.63) | 66.42 (6.82) | 50.80 (18.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7 | 8 | 9 | 8 | 9 | 6 | 54
  Male | 9 | 8 | 5 | 4 | 3 | 4 | 3 | 6 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 96
Weight [Mean (Standard Deviation); unit: kg] | 72.74 (11.43) | 71.68 (11.67) | 71.40 (14.40) | 71.02 (13.80) | 76.05 (11.88) | 70.90 (10.69) | 69.06 (14.25) | 84.43 (17.53) | 73.41 (13.66)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.89 (2.92) | 24.23 (3.68) | 23.80 (2.74) | 23.69 (2.03) | 25.92 (1.66) | 24.69 (3.09) | 24.03 (3.17) | 26.73 (2.75) | 24.62 (2.91)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactions at the Injection Site (Pain, Tenderness, Erythema/Redness, Induration/Swelling) Recorded up to 7 Days After Each IMP Dose
Description: Solicited local reactions at the injection site (pain, tenderness, erythema/redness, and induration/swelling) were monitored and graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". The reporting of local reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
Time Frame: From Day 1 to Day 8 for Prime Immunization and from Day 22 to Day 29 for Boost Immunization
Population: Safety Set - All participants who received at least one dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Prime up to Day 7 after Prime: Number of participants with any local reaction: number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  Prime up to Day 7 after Prime: Number of participants with any local reaction | 9 | 9 | 12 | 12 | 4 | 10 | 10 | 9
  Prime up to Day 7 after Prime: Number of participants with any grade >= 3 local reaction: number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  Prime up to Day 7 after Prime: Number of participants with any grade >= 3 local reaction | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any local reaction: number analyzed (Participants) | 12 | 12 | 12 | 0 | 12 | 11 | 12 | 12
  Boost up to Day 7 after Boost: Number of participants with any local reaction | 9 | 9 | 12 |  | 2 | 9 | 8 | 11
  Boost up to Day 7 after Boost: Number of participants with any grade >= 3 local reaction: number analyzed (Participants) | 12 | 12 | 12 | 0 | 12 | 11 | 12 | 12
  Boost up to Day 7 after Boost: Number of participants with any grade >= 3 local reaction | 0 | 0 | 1 |  | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Systemic Reactions (Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, Arthralgia, Chills, Loss of Appetite, Malaise, and Fever) Recorded up to 7 Days After Each IMP Dose
Description: Solicited systemic reactions (nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever) were monitored and graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". The reporting of systemic reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
Time Frame: From Day 1 to Day 8 for Prime Immunization and from Day 22 to Day 29 for Boost Immunization
Population: Safety Set - All participants who received at least one dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Prime up to Day 7 after Prime: Number of participants with any systemic reaction: number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  Prime up to Day 7 after Prime: Number of participants with any systemic reaction | 4 | 10 | 12 | 12 | 3 | 9 | 9 | 10
  Prime up to Day 7 after Prime: Number of participants with any grade >= 3 systemic reaction: number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  Prime up to Day 7 after Prime: Number of participants with any grade >= 3 systemic reaction | 0 | 0 | 1 | 3 | 0 | 3 | 0 | 2
  Boost up to Day 7 after Boost: Number of participants with any systemic reaction: number analyzed (Participants) | 12 | 12 | 12 | 0 | 12 | 11 | 12 | 12
  Boost up to Day 7 after Boost: Number of participants with any systemic reaction | 10 | 9 | 12 |  | 2 | 10 | 9 | 12
  Boost up to Day 7 after Boost: Number of participants with any grade >= 3 systemic reaction: number analyzed (Participants) | 12 | 12 | 12 | 0 | 12 | 11 | 12 | 12
  Boost up to Day 7 after Boost: Number of participants with any grade >= 3 systemic reaction | 0 | 2 | 4 |  | 0 | 2 | 2 | 2

3. Primary Outcome: The Percentage of Participants With at Least 1 Unsolicited Treatment Emergent Adverse Event (TEAE) Occurring After Prime Immunization up to Boost Immunization or 28 Days After Prime Immunization
Description: Treatment emergent adverse events (TEAEs) were analyzed by age group, dose level, and for each IMP dose. The number and percentage of participants reporting at least one TEAE was summarized by adverse event types (any TEAE and any grade >=3 TEAE) using the Safety Set.
Time Frame: 28 days following first IMP dose or up to second IMP dose (whichever was first)
Population: Safety Set - All participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
percentage of participants
  Any TEAE | 42 | 25 | 25 | 50 | 17 | 17 | 25 | 42
  Any grade >=3 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: The Percentage of Participants With at Least 1 Unsolicited TEAE Occurring up to 28 Days After Boost Immunization or After Prime Immunization (if no Boost Immunization)
Description: Treatment emergent adverse events (TEAEs) were analyzed by age group, dose level, and for each IMP dose. The percentage of participants reporting at least one TEAE was summarized by adverse event types (any TEAE and any grade >=3 TEAE) using the Safety Set.
Time Frame: 28 days following second IMP dose or first IMP dose (if no second IMP dose as given)
Population: Safety Set - All participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
percentage of participants
  Any TEAE | 50 | 33 | 42 | 50 | 58 | 25 | 42 | 50
  Any grade >=3 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8

5. Secondary Outcome: Functional Antibody Responses
Description: At 7 and 21 days after primary immunization and at 7, 14, 21, 28 days after boost immunization.
Time Frame: up to 50 days following first IMP dose
Population: Immunogenicity set - all participants who received at least one dose of IMP and had at least one post-baseline functional antibody titer immunogenicity assessment.
  Boost immunization withheld for 30 μg younger cohort following Safety Review Committee decision.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
titer
  7 days after Prime Immunization (Day 8) | 5.0 [5.0 to 5.0] | 5.1 [4.8 to 5.5] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 7.3 [3.2 to 16.6] | 5.0 [5.0 to 5.0]
  21 days after Prime Immunization (Day 22) | 6.1 [4.5 to 8.4] | 25.9 [13.8 to 48.7] | 8.9 [6.0 to 13.3] | 12.2 [7.5 to 20.0] | 6.3 [4.8 to 8.3] | 5.3 [4.9 to 5.8] | 15.0 [5.9 to 37.9] | 9.4 [5.4 to 16.4]
  7 days after Boost Immunization (Day 29) | 51.5 [26.4 to 100.3] | 479.5 [300.3 to 765.5] | 106.8 [58.2 to 196.0] | 10.0 [6.5 to 15.4] | 53.4 [25.1 to 113.7] | 51.9 [25.0 to 107.4] | 320.0 [189.7 to 539.7] | 207.5 [118.0 to 364.8]
  14 days after Boost Immunization (Day 36) | 60.6 [33.5 to 109.8] | NA [NA to NA] — Missing Day 36 data of 10 μg younger cohort as they have only re-consented to Clinical Trial Protocol 7.0 (introducing visit 5a/Day 36) on/after their Day 43. | NA [NA to NA] — Missing Day 36 data of 20 μg younger cohort as they have only re-consented to Clinical Trial Protocol 7.0 (introducing visit 5a/Day 36) on/after their Day 43. | 10.3 [6.9 to 15.4] | 77.7 [40.4 to 149.4] | 219.8 [148.5 to 325.4] | 320.0 [169.3 to 604.9] | 359.2 [204.0 to 632.6]
  21 days after Boost Immunization (Day 43) | 36.4 [20.0 to 66.2] | 116.5 [79.6 to 170.4] | 201.6 [104.9 to 387.2] | 9.7 [5.7 to 16.5] | 53.4 [27.5 to 103.6] | 155.4 [105.0 to 230.1] | 285.1 [152.6 to 532.7] | 261.4 [136.0 to 502.6]
  28 days after Boost Immunization (Day 50) | 31.7 [18.5 to 54.6] | 80.0 [49.1 to 130.4] | 219.8 [117.5 to 411.1] | 7.9 [5.0 to 12.5] | 41.2 [20.5 to 82.8] | 138.5 [87.9 to 218.2] | 232.9 [131.1 to 413.8] | 195.8 [109.4 to 350.6]

6. Secondary Outcome: Fold Increase in Functional Antibody Titers
Description: At 7 and 21 days after primary immunization and at 7, 14, 21, and 28 days after the boost immunization.
Time Frame: up to 50 days following first IMP dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Fold rise
  7 days after Prime Immunization (Day 8) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.3 [0.8 to 2.1] | 1.0 [1.0 to 1.0]
  21 days after Prime Immunization (Day 22) | 1.2 [0.9 to 1.7] | 5.2 [2.8 to 9.7] | 1.8 [1.2 to 2.7] | 2.4 [1.5 to 4.0] | 1.3 [1.0 to 1.7] | 1.1 [1.0 to 1.2] | 2.6 [1.3 to 5.0] | 1.9 [1.1 to 3.3]
  7 days after Boost Immunization (Day 29): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  7 days after Boost Immunization (Day 29) | 10.3 [5.3 to 20.1] | 95.9 [60.1 to 153.1] | 21.4 [11.6 to 39.2] | 2.0 [1.3 to 3.1] | 10.7 [5.0 to 22.7] | 10.4 [5.0 to 21.5] | 55.4 [35.5 to 86.4] | 41.5 [23.6 to 73.0]
  14 days after Boost Immunization (Day 36): number analyzed (Participants) | 10 | 0 | 0 | 12 | 12 | 12 | 12 | 12
  14 days after Boost Immunization (Day 36) | 12.1 [6.7 to 22.0] |  |  | 2.1 [1.4 to 3.1] | 15.5 [8.1 to 29.9] | 44.0 [29.7 to 65.1] | 55.4 [31.2 to 98.4] | 71.8 [40.8 to 126.5]
  21 days after Boost Immunization (Day 43): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  21 days after Boost Immunization (Day 43) | 7.3 [4.0 to 13.2] | 23.3 [15.9 to 34.1] | 40.3 [21.0 to 77.4] | 1.9 [1.1 to 3.3] | 10.7 [5.5 to 20.7] | 31.1 [21.0 to 46.0] | 49.4 [29.7 to 81.9] | 52.3 [27.2 to 100.5]
  28 days after Boost Immunization (Day 50): number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  28 days after Boost Immunization (Day 50) | 6.3 [3.7 to 10.9] | 16.0 [9.8 to 26.1] | 44.0 [23.5 to 82.2] | 1.6 [1.0 to 2.5] | 8.2 [4.1 to 16.6] | 27.7 [17.6 to 43.6] | 40.3 [26.7 to 60.9] | 39.2 [21.9 to 70.1]

7. Secondary Outcome: Number of Participants With Seroconversion Defined as a Minimum of 4-fold Increase of Functional Antibody Titers as Compared to Baseline
Description: At 7 and 21 days after primary immunization and at 7, 14, 21, and 28 days after the boost immunization.
Time Frame: up to 50 days following first IMP dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  7 days after Prime Immunization (Day 8) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  21 days after Prime Immunization (Day 22) | 1 | 9 | 2 | 5 | 1 | 0 | 4 | 2
  7 days after Boost Immunization (Day 29): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  7 days after Boost Immunization (Day 29) | 9 | 12 | 12 | 3 | 10 | 10 | 12 | 12
  14 days after Boost Immunization (Day 36): number analyzed (Participants) | 10 | 0 | 0 | 12 | 12 | 12 | 12 | 12
  14 days after Boost Immunization (Day 36) | 9 |  |  | 4 | 11 | 12 | 12 | 12
  21 days after Boost Immunization (Day 43): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  21 days after Boost Immunization (Day 43) | 8 | 12 | 12 | 3 | 9 | 12 | 12 | 12
  28 days after Boost Immunization (Day 50): number analyzed (Participants) | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12
  28 days after Boost Immunization (Day 50) | 8 | 11 | 12 | 1 | 9 | 12 | 12 | 12

8. Secondary Outcome: Functional Antibody Responses
Description: At 63, 162, 365 days after boost immunization.
Time Frame: From 51 to up to 387 days following first IMP dose
Population: Immunogenicity set - all participants who received at least one dose of IMP and had at least one post-baseline functional antibody titer immunogenicity assessment.
  Boost immunization withheld for 30 μg younger cohort following Safety Review Committee decision.
  Day 387 (365 days after boost) data is either missing due to exclusion because of non-study vaccination or due to premature discontinuation.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
titer
  63 days after Boost Immunization (Day 85): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 12
  63 days after Boost Immunization (Day 85) | 40.0 [22.4 to 71.4] | 51.9 [39.1 to 68.9] | 116.5 [51.0 to 266.1] | 13.0 [7.8 to 21.5] | 34.6 [18.1 to 66.1] | 85.2 [48.7 to 149.0] | 142.5 [77.9 to 260.7] | 75.5 [45.6 to 125.0]
  162 days after Boost Immunization (Day 184): number analyzed (Participants) | 11 | 11 | 12 | 11 | 8 | 8 | 6 | 7
  162 days after Boost Immunization (Day 184) | 11.7 [5.8 to 23.8] | 51.5 [33.9 to 78.1] | 119.9 [62.6 to 229.5] | 11.0 [4.7 to 25.8] | 9.6 [6.1 to 15.0] | 28.3 [11.2 to 71.6] | 44.9 [22.0 to 91.8] | 107.7 [42.3 to 273.8]
  365 days after Boost Immunization (Day 387): number analyzed (Participants) | 5 | 5 | 11 | 1 | 1 | 0 | 0 | 0
  365 days after Boost Immunization (Day 387) | 197.0 [14.2 to 2727.9] | 452.5 [47.4 to 4322.3] | 513.3 [215.8 to 1221.2] | 5.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available | 1280.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available |  |  |

9. Secondary Outcome: Fold Increase in Functional Antibody Titers
Description: At 63, 162, 365 days after boost immunization.
Time Frame: From 51 to up to 387 days following first IMP dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Fold rise
  63 days after Boost Immunization (Day 85): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 12
  63 days after Boost Immunization (Day 85) | 8.0 [4.5 to 14.3] | 10.4 [7.8 to 13.8] | 23.3 [10.2 to 53.2] | 2.6 [1.6 to 4.3] | 6.9 [3.6 to 13.2] | 17.0 [9.7 to 29.8] | 24.7 [15.3 to 39.9] | 15.1 [9.1 to 25.0]
  162 days after Boost Immunization (Day 184): number analyzed (Participants) | 11 | 11 | 12 | 11 | 8 | 8 | 6 | 7
  162 days after Boost Immunization (Day 184) | 2.3 [1.2 to 4.8] | 10.3 [6.8 to 15.6] | 24.0 [12.5 to 45.9] | 2.2 [0.9 to 5.2] | 1.9 [1.2 to 3.0] | 5.7 [2.2 to 14.3] | 9.0 [4.4 to 18.4] | 21.5 [8.5 to 54.8]
  365 days after Boost Immunization (Day 387): number analyzed (Participants) | 5 | 5 | 11 | 1 | 1 | 0 | 0 | 0
  365 days after Boost Immunization (Day 387) | 39.4 [2.8 to 545.6] | 90.5 [9.5 to 864.5] | 102.7 [43.2 to 244.2] | 1.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available | 256.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available |  |  |

10. Secondary Outcome: Number of Participants With Seroconversion Defined as a Minimum of 4-fold Increase of Functional Antibody Titers as Compared to Baseline
Description: At 63, 162, 365 days after boost immunization.
Time Frame: From 51 to up to 387 days following first IMP dose
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  63 days after Boost Immunization (Day 85): number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 12
  63 days after Boost Immunization (Day 85) | 9 | 12 | 11 | 3 | 8 | 11 | 12 | 12
  162 days after Boost Immunization (Day 184): number analyzed (Participants) | 11 | 11 | 12 | 11 | 8 | 8 | 6 | 7
  162 days after Boost Immunization (Day 184) | 4 | 11 | 12 | 2 | 2 | 6 | 6 | 6
  365 days after Boost Immunization (Day 387): number analyzed (Participants) | 5 | 5 | 11 | 1 | 1 | 0 | 0 | 0
  365 days after Boost Immunization (Day 387) | 4 | 5 | 11 | 0 | 1 |  |  |

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events: within 7 days after each IMP dose; SAEs: from Day 1 (Dose 1 [Prime Immunization]) up to Day 387 (approximately 12 months after Dose 2 [Boost Immunization]); Other AEs in participants with Dose 2: All AEs from Day 1 up to Day 50 and in addition if assessed as IMP-related from Day 50 up to Day 387; Other AEs in participants without Dose 2: All AEs from Day 1 up to Day 29 and in addition if assessed as IMP-related from Day 29 up to Day 387.
Arm/Group | Part A Participants Aged 18 to 55 Years - 3 μg | Part A Participants Aged 18 to 55 Years - 10 μg | Part A Participants Aged 18 to 55 Years - 20 μg | Part A Participants Aged 18 to 55 Years - 30 μg | Part A Participants Aged 56 to 85 Years - 3 μg | Part A Participants Aged 56 to 85 Years - 10 μg | Part A Participants Aged 56 to 85 Years - 20 μg | Part A Participants Aged 56 to 85 Years - 30 μg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 1/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 4/12 | 5/12 | 6/12 | 7/12 | 5/12 | 5/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | Part A Participants Aged 56 to 85 Years - 3 μg (N=12) | Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | Part A Participants Aged 56 to 85 Years - 30 μg (N=12)
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | Part A Participants Aged 56 to 85 Years - 3 μg (N=12) | Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | Part A Participants Aged 56 to 85 Years - 30 μg (N=12)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 3 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental care (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04537949/Prot_002.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT04537949/SAP_003.pdf